CLINICAL TRIAL: NCT02428868
Title: Use of Combined Tranexamic Acid and Intravenous Iron for Hip Fracture Surgery in Elderly
Brief Title: IV Iron in Association With Tranexamic Acid for Hip Fracture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Institut Kassab d'Orthopédie (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: P-2015004/AR
Record Dates: First submitted 2015-04-14; First posted 2015-04-29 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2015-04

CONDITIONS: Hip Fracture; Anemia
Keywords: hip fracture; anemia; blood transfusion; tranexamic acid; intravenous iron
MeSH Terms: conditions — Hip Fractures; Anemia | interventions — Tranexamic Acid; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Tranexamic acid - intravenous iron (Experimental): IV iron (Ferroven®) : 2 vials of 10 mL containing each one 100 mg iron, diluted in 100 mL normal saline over 30 minutes before induction of anesthesia and repeated on day two and three.
  IV Tranexamic acid (Exacyl®): 1 gram diluted in 20 mL saline solution, in 30 minutes, five minutes before skin incision and a second 1 gram, 3 hours later.
  Interventions: Drug: tranexamic acid (Exacyl®); Drug: intravenous iron (Ferroven®)
- Tranexamic acid (Active Comparator): IV Tranexamic acid (Exacyl®): 1 gram diluted in 20 mL saline solution, in 30 minutes, five minutes before skin incision and a second 1 gram, 3 hours later.
  Interventions: Drug: tranexamic acid (Exacyl®)
- Placebo (Placebo Comparator): 20 mL saline, in 30 minutes, five minutes before skin incision and 20 ml 3 hours later.
  Interventions: Other: Saline

INTERVENTIONS:
Drug: tranexamic acid (Exacyl®) — 1 gram diluted in 20 mL saline solution, in 30 minutes, five minutes before skin incision and a second 1 gram, 3 hours later
  Arms: Tranexamic acid; Tranexamic acid - intravenous iron
Drug: intravenous iron (Ferroven®) — 2 vials of 10 mL containing each one 100 mg iron, diluted in 100 mL normal saline over 30 minutes before induction of anesthesia and repeated on day two and three.
  Arms: Tranexamic acid - intravenous iron
Other: Saline — 20 mL saline in 30 minutes, five minutes before skin incision and 20 ml 3 hours later.
  Arms: Placebo

SUMMARY:
It is a prospective randomized controlled study aiming to test if tranexamic acid combined to intravenous iron before and after surgery for hip fracture in elderly can decrease peri-operative red cell transfusion.

DETAILED DESCRIPTION:
Hip fracture is an increasing problem. Anemia is a common finding in these patients with a prevalence ranging from 24% to 44% and is a strong negative prognostic marker. Several studies have explored whether interventions to improve anemia result in better outcomes. Thus, alternatives to allogenic red cell transfusion have been suggested in hip fracture, such as IV iron and tranexamic acid.

The aim of the study is to test the effect of combination of IV iron with tranexamic acid before and after surgery for hip fracture on incidence of peri-operative red cell transfusion.

It is a prospective randomized single-blinded monocentric study including 150 patients undergoing hip fracture surgery within 72 h after trauma aged ≥ 60 years divided in 3 groups: Group A (IV fer+Tranexamic acid), Group B (Tranexamic acid), Group C (placebo). The main outcome was percentage of patients who receive red-cell transfusion during hospitalization. Hemoglobin levels up to 60 days post-operatively and incidence of thrombotic events were secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing hip fracture surgery within 72 h after trauma.

Exclusion Criteria:

* Vascular events within the last 2 months such as cerebrovascular accident (CVA), Myocardial infarction (MI), Venous Thromboembolism (VTE) and/or recurrent VTE or arterial thrombosis.
* Patients receiving anticoagulation therapy with warfarin or clopidogrel.
* History of seizures.
* Multiple fractures.
* Transfusion received during admission, prior to surgery (Hb< 8g/dl).
* Creatinine clearance less than 30 mL/min
* Known history of Factor V Leiden, protein C/S deficiency, prothrombin gene mutation, anti-thrombin deficiency, anti-phospholipid antibody syndrome, lupus anticoagulant
* Coronary stent placement within the previous 6 months
* Disseminated intravascular coagulation
* Subarachnoid hemorrhage
* Allergy for tranexamic acid
* Hypersensitivity to Iron sucrose or any component of the formulation
* Clinical signs of acute thromboembolic event
* Malignancy
* Body weight > 100kg
* Advanced Dementia

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2015-04; Primary Completion 2016-04 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
transfusion | 5 days
  percentage of patients who receive red-cell transfusion during hospitalization

SECONDARY OUTCOMES:
Average red-cell packs per patient | 5 days
blood loss | 5 days
  Calculated blood loss per patient from admission to day 5 postoperatively
haemoglobin level | day 1
  haemoglobin level at day 1 postoperatively
haemoglobin level | day 2
haemoglobin level | day 5
haemoglobin level | day 30
haemoglobin level | day 60
Thromboembolic events | day 60
  stroke or transient ischemic attack, venous thromboembolism and clinically recognized myocardial during hospital stay and until 60 days postoperatively.
Post-operative bacterial infection | day 60
  urinary tract infection, lower respiratory tract infection, pneumonia and superficial or deep wound infection.
number of days in hospital | day 10
  expected period of approximately 5 days
Functional mobility | day 60
  ability to walk more than 10 m or outside home 60 days after hospital discharge.
mortality | 5 days
  in-hospital mortality
mortality | day 30
mortality | day 60

CONTACTS AND LOCATIONS:
Overall Officials: Olfa Kaabachi, Professor, Principal Investigator — Institut Mohamed Kassab d'Orthopédie
Locations (1):
- Institut Mohamed Kassab d'Orthopédie, Manouba, La Manouba, Tunisia

REFERENCES:
- [Background] Hagino T, Ochiai S, Sato E, Maekawa S, Wako M, Haro H. The relationship between anemia at admission and outcome in patients older than 60 years with hip fracture. J Orthop Traumatol. 2009 Sep;10(3):119-22. doi: 10.1007/s10195-009-0060-8. Epub 2009 Aug 26. PMID 19707842
- [Background] Carson JL, Terrin ML, Noveck H, Sanders DW, Chaitman BR, Rhoads GG, Nemo G, Dragert K, Beaupre L, Hildebrand K, Macaulay W, Lewis C, Cook DR, Dobbin G, Zakriya KJ, Apple FS, Horney RA, Magaziner J; FOCUS Investigators. Liberal or restrictive transfusion in high-risk patients after hip surgery. N Engl J Med. 2011 Dec 29;365(26):2453-62. doi: 10.1056/NEJMoa1012452. Epub 2011 Dec 14. PMID 22168590
- [Result] Spahn DR. Anemia and patient blood management in hip and knee surgery: a systematic review of the literature. Anesthesiology. 2010 Aug;113(2):482-95. doi: 10.1097/ALN.0b013e3181e08e97. PMID 20613475
- [Result] Serrano-Trenas JA, Ugalde PF, Cabello LM, Chofles LC, Lazaro PS, Benitez PC. Role of perioperative intravenous iron therapy in elderly hip fracture patients: a single-center randomized controlled trial. Transfusion. 2011 Jan;51(1):97-104. doi: 10.1111/j.1537-2995.2010.02769.x. PMID 20630042
- [Result] Zufferey PJ, Miquet M, Quenet S, Martin P, Adam P, Albaladejo P, Mismetti P, Molliex S; tranexamic acid in hip-fracture surgery (THIF) study. Tranexamic acid in hip fracture surgery: a randomized controlled trial. Br J Anaesth. 2010 Jan;104(1):23-30. doi: 10.1093/bja/aep314. PMID 19926634